CLINICAL TRIAL: NCT06079333
Title: NEO- and Adjuvant Targeted Therapy in Braf-mutated Anaplastic Cancer of the Thyroid (NEO-ATACT Study)
Acronym: NEO-ATACT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, HW Kapiteijn, MD, PhD, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEOAC
Record Dates: First submitted 2023-06-29; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Anaplastic Thyroid Cancer
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — dabrafenib; trametinib

STUDY DESIGN:
Intervention Model Description: prospective, non-randomized, single center, open-label phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- neo-adjuvant and adjuvant braf/mek-inhibition (Experimental): Participants will undergo neo-adjuvant treatment with dabrafenib/trametinib. After 6 weeks of BRAF/MEK inhibitors, participants will undergo an evaluation of resectability. If the tumor is resectable, patients undergo tumor resection. If not resectable, neo-adjuvant treatment continues for another 6 weeks followed by a new evaluation. All resected patients receive adjuvant dabrafenib/trametinib up to a total treatment duration of 52 weeks. If resection is not possible, patients will continue on dabrafenib/trametinib.
  Interventions: Drug: dabrafenib/trametinib

INTERVENTIONS:
Drug: dabrafenib/trametinib — braf/mek-inhibition

SUMMARY:
Anaplastic thyroid cancer (ATC) is an almost invariable lethal cancer in humans.

Most patients present with a rapid progressive mass in the neck with progressive complaints like dyspnoea, dysphagia or pain. The risk of suffocation is the main reason for rapid surgical intervention, but we know from literature that an oncological resection with clear margins is seldomly achieved. Some patients deteriorate that fast after surgery that radiation therapy and/or chemotherapy is not feasible anymore. Patients with BRAF-mutated ATC already have shown to benefit from targeted BRAF/MEK inhibition. This study aims to increase the number of patients that undergo a successful R0 tumor resection after neo-adjuvant BRAF/MEK inhibitor treatment.

DETAILED DESCRIPTION:
Unmet need ATC is a very serious condition and is, apart from a few exclusive cases, always lethal. Many patients suffer uncontrollable loco-regional disease with even so uncontrollable complaints of airway obstruction, oesophagus obstruction, pain and neck movement impairment. One of the only shown beneficial treatment is complete surgical resection with clear surgical margins combined with radiotherapy and systemic treatment. However, in less than 10-15% of the patients the pathologist reports clear surgical margins. Thereby it is noticeable that surgery often results in serious morbidity, due to an esophagectomy, laryngectomy or trachea resection all accompanied by an extensive reconstruction. All of these come with serious morbidity and seldomly lead to clear margins and better outcome.

Proposed solution A single center, phase II study for the evaluation of safety and efficacy of neo-adjuvant and adjuvant dabrafenib/trametinib treatment in BRAF mutated ATC patients. By introducing neo-adjuvant treatment the hypothesis is that better selection is done for patients who are eligible for complete surgery and that surgery results more often in clear surgical margins after neo-adjuvant treatment. Second benefit of treating patients with combined loco-regional and systemic agents before surgery is that micro/macrometastases (being there in at least 30% of the patients at diagnosis) are already being treated directly after diagnosis. Lastly, adjuvant treatment with dabrafenib/trametinib will hopefully result in reduction of local and distant recurrences after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. Age over 18 years old.
3. World Health Organization (WHO) Performance Status 0 or I.
4. Histologically confirmed ATC (centrally reviewed).
5. Confirmed presence of BRAFV600E/K mutation in primary tumor tissue.
6. No distant metastases (M0).
7. Free or secured airway.
8. Able to swallow pills.
9. Patients must have undergone complete disease staging including: PET-CT scan and CT-neck/thorax/abdomen.
10. No prior anticancer systemic treatment (including chemotherapy, immunotherapy, oncolytic viral therapy, other systemic therapies).
11. No prior radiotherapy to site of interest.
12. Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Neutrophils ≥ 1.0x109/L, Platelets ≥ 100 x109/L, Hemoglobin ≥ 6.5 mmol/L, AST ≤ 2.5 x ULN, ALT ≤ 2.5 x ULN, Total bilirubin ≤ 1.5 X ULN, INR and PTT in normal range, LDH < 2xULN. Serum creatinine ≤ 1.5 × ULN; or calculated creatinine clearance ≥ 50 mL/min by Cockcroft-Gault formula; or estimated glomerular filtration rate > 50 mL/min/1.73m2.
13. Absence of additional severe and/or uncontrolled concurrent disease.

Exclusion Criteria:

1. No informed consent.
2. History of cancer within 2 years from diagnosis of ATC (exception: basal cell skin cancer, in situ carcinoma).
3. Poorly differentiated transformation of previous differentiated thyroid cancer.
4. Presence of distant metastases.
5. Underlying medical conditions that, in the Investigator's opinion, will make the administration of study treatment hazardous or obscure the interpretation of toxicity determination or adverse events
6. History of congestive heart failure, active cardiac conditions, including unstable coronary syndromes, significant arrhythmias and severe valvular disease must be evaluated for risks of undergoing general anesthesia.
7. Pregnancy or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
primary endpoint of the study will be R0 resection rate (efficacy). | after 6-12 weeks braf/mek-inhibition
  primary endpoint of the study will be R0 resection rate (efficacy).

SECONDARY OUTCOMES:
Neo-adjuvant and adjuvant treatment related toxicity of dabrafenib/trametinib (according to CTCAE v. 5.0) | during 1 year of treatment with braf/mek-inhibition
  Neo-adjuvant and adjuvant treatment related toxicity of dabrafenib/trametinib (according to CTCAE v. 5.0) during 1 year of treatment with braf/mek-inhibition
30-day postoperative surgical complications | within 30 days after surgery
  30-day postoperative surgical complications (within 30 days after surgery)
Histopathological response after neo-adjuvant treatment | 6-12 weeks neo-adjuvant braf/mek-inhibition
  Histopathological response after neo-adjuvant treatment: complete response (<10% tumor cells), partial response (between more than 10% and up to 50% tumor cells), or no response (still more than 50% tumor cells)
Locoregional-free survival | at 2 years
  Locoregional-free survival
Distant metastasis-free survival | at 2 years
  Distant metastasis-free survival
Overall survival | at 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Kapiteijn, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Ellen Kapiteijn, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No